CLINICAL TRIAL: NCT04434963
Title: Safety and Feasibility of Reversible Induction Strategy Supported by HFNC Combined With Specific Anesthetic
Brief Title: Safety and Feasibility of Reversible Induction Strategy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, diansan su, Principal Investigator, RenJi Hospital
Other Study IDs: RenjiH6502
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Patients With Uncertain Difficult Airway; Colon Cancer; Gastric Cancer; Prostatic Cancer
Keywords: THRIVE; Uncertain difficult airway; Reversible induction strategy
MeSH Terms: conditions — Colonic Neoplasms; Stomach Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study would explore the safety and feasibility of a reversible induction strategy for uncertain difficult airway. This reversible induction strategy would include high flow nasal canular oxygenation support, short-term effect anesthetic including Propofol and Remifentanil for sedation and analgesia and Sugammadex would be used for reverse the muscle relaxant.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old,<65 years old
* Signed informed consent
* Undergoing selective operation （ time of operation is over two hours）
* ASA classification I-II
* Mallampati classification 3-4
* suspicious difficult airway, but the anesthetists decide to try to rapid induction

Exclusion Criteria:

* Patients with several dysfunctions of liver, kidney or heart)
* Patients with a full stomach or have other risk factors of reflux aspiration
* Any medicine was taken before surgery, which might enhance or mitigate the effects of muscle relaxant
* Infection of the mouth or nose
* Allergy history of any medicine which would be used in this study
* Pregnant and lactating women
* Patients with neuromuscular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an uncertain difficult airway, who will undergo a selective operation and need trachea intubtion.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Successful rate of reversion | From the beginning of induction to 15min later

SECONDARY OUTCOMES:
TOFr 0.9 reversion time | From the beginning of induction to 15min later
BIS 80 reversion time | From the beginning of induction to 15min later
Tidal volume 6-8ml tidal volume 6-8ml/kg reversion time | From the beginning of induction to 15min later
consciousness reversion time | From the beginning of induction to 15min later

CONTACTS AND LOCATIONS:
Overall Officials: diansan su, Study Director — Renji Hospital, Shanghai Jiaotong University, Shanghai, China
Locations (1):
- Ren Ji Hospital Affliated to School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
IPD is unavailable to other researchers